CLINICAL TRIAL: NCT05002972
Title: Tanglewood Trail Walking Program to Increase Phytonutrient Intake and Physical Activity in a Rural Kentucky Town
Brief Title: Tanglewood Trail Walking Program in Rural Kentucky 2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dawn Brewer (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Dawn Brewer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-0283-P2H 2019; P42ES007380 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Dietary Habits
Keywords: farmers market; Appalachia; physical activity; fruit and vegetable voucher program
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking Group (Experimental): Subjects will participate in a walking group led by a community organizer as a means to get to a local farmer's market.
  Interventions: Behavioral: walking group led by a community organizer

INTERVENTIONS:
Behavioral: walking group led by a community organizer — Subjects will walk 1 kilometer from a pre-determined point to a local farmer's market.

SUMMARY:
The Tanglewood Trail Walking Program is a well established community health initiative that encourages community members to walk approximately 1 mile to the Whitesburg Farmers Market each Saturday. The study aims to determine if walking to the market with a community health coach results in healthier options being selected at the market when compared to the driving group.

DETAILED DESCRIPTION:
In the summer of 2017, community members of Whitesburg, KY were recruited to join the Tanglewood Trail Walking Program to the Whitesburg farmers market. Each Saturday, participants reported whether or not they walked the 1 mile trail to the farmers market and they reported which fruits and vegetables they purchased. Participants completed questionnaires about fruit and vegetable consumption and physical activity. Participants also provided physical and biological measurements. The ClinicalTrials.gov record for the original trial in 2017 is NCT03495648.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk 1 kilometer

Exclusion Criteria:

* pregnant
* institutionalized adults
* impaired consent ability
* prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Brewer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Walking Group
Started | 63
Completed | 61
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Walking Group
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 55
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Carotenoid Levels
Description: Subjects' carotenoid status will be measured using a carotenoid Raman Spectroscopy to determine if walking combined with a voucher for fruits and vegetables increases intake in fruits and vegetables as measured by carotenoid status.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: relative units (absorbance)
Arm/Group | Walking Group
Number analyzed (Participants) | 63
relative units (absorbance)
  baseline | 148.7 (65.7)
  post-study: number analyzed (Participants) | 53
  post-study | 176.4 (69.3)

2. Primary Outcome: Self-reported Fruit Intake
Description: Subjects' self-reported fruit intake will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant self-reported fruit intake.
Time Frame: 3 months
Population: Not all participants completed this outcome measure
Measure: Mean (Standard Deviation); unit: servings of fruit per day
Arm/Group | Walking Group
Number analyzed (Participants) | 62
servings of fruit per day
  baseline | 1.8 (1.6)
  post-study | 1.7 (1.2)

3. Primary Outcome: Self-reported Vegetable Intake
Description: Subjects' self-reported vegetable intake will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant self-reported vegetable intake.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: servings of vegetables per day
Arm/Group | Walking Group
Number analyzed (Participants) | 62
servings of vegetables per day
  baseline | 4.2 (2.6)
  post-study: number analyzed (Participants) | 56
  post-study | 4.1 (2.3)

4. Secondary Outcome: A1c Levels
Description: Subjects' A1c will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant A1c.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Walking Group
Number analyzed (Participants) | 61
percentage of glycated hemoglobin
  baseline | 5.6 (0.7)
  post-study: number analyzed (Participants) | 55
  post-study | 5.4 (0.9)

5. Secondary Outcome: LDL Cholesterol Levels
Description: Subjects' LDL will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant LDL.
Time Frame: 3 months
Population: Not all participants completed this study outcome.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Walking Group
Number analyzed (Participants) | 46
mg/dl
  baseline: number analyzed (Participants) | 45
  baseline | 83.8 (31.8)
  post-study | 85.9 (29.3)

6. Secondary Outcome: HDL Cholesterol Levels
Description: Subjects' HDL will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant HDL
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Walking Group
Number analyzed (Participants) | 56
mg/dl
  baseline | 47.3 (10.5)
  post-study: number analyzed (Participants) | 51
  post-study | 46.4 (11.1)

7. Secondary Outcome: Total Cholesterol Levels
Description: Subjects' total cholesterol will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant total cholesterol.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Walking Group
Number analyzed (Participants) | 60
mg/dl
  baseline | 161.8 (34.9)
  post-study: number analyzed (Participants) | 54
  post-study | 170.8 (35.3)

8. Secondary Outcome: Weight
Description: Subjects' weight will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant weight.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Walking Group
Number analyzed (Participants) | 63
pounds
  baseline | 205.3 (61.6)
  post-study: number analyzed (Participants) | 55
  post-study | 207.8 (61.0)

9. Secondary Outcome: Waist Circumference
Description: Subjects' waist circumference will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant waist circumference.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Walking Group
Number analyzed (Participants) | 47
inches
  baseline | 42.9 (8.5)
  post-study | 43.1 (8.3)

10. Secondary Outcome: Hours of Vigorous Exercise
Description: Subjects will self-report the number of hours spent in vigorous exercise per week.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Walking Group
Number analyzed (Participants) | 52
hours per week
  baseline | 2.2 (2.0)
  post-study: number analyzed (Participants) | 32
  post-study | 3.54 (7.21)

11. Secondary Outcome: Hours of Moderate Exercise
Description: Subjects will self-report the number of hours spent in moderate exercise per week.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Walking Group
Number analyzed (Participants) | 54
hours per week
  baseline | 4.6 (11.1)
  post-study | 2.4 (2.1)

12. Secondary Outcome: Hours of Sitting
Description: Subjects will self-report the number of hours spent sitting per day.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Walking Group
Number analyzed (Participants) | 58
hours per week
  baseline | 6.0 (6.1)
  post-study: number analyzed (Participants) | 56
  post-study | 4.6 (2.9)

13. Secondary Outcome: Hours of Walking Per Week
Description: Subjects will self-report the number of hours spent walking per week.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Walking Group
Number analyzed (Participants) | 58
hours per week
  baseline | 3.0 (6.4)
  post-study | 3.8 (12.3)

14. Secondary Outcome: Understanding of Plant-based Phytonutrients
Description: Participants will be asked a question demonstrating their understanding of the importance of ingesting plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 62
Participants
  baseline | 42
  post-study: number analyzed (Participants) | 55
  post-study | 42

15. Secondary Outcome: Belief in the Benefit of Plant-based Nutrients
Description: Participants will be asked a question demonstrating their appreciation of plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 42
Participants
  baseline | 41
  post-study | 40

16. Secondary Outcome: Belief in the Preventative Effects of Plant-Based Nutrients
Description: Participants will be asked a question demonstrating their beliefs of plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 42
Participants
  baseline | 38
  post-study | 7

17. Secondary Outcome: Belief in the Role of Healthy Diet in Protecting Health From Pollutants
Description: Participants will be asked a question demonstrating their beliefs that a healthy diet might protect health from environmental pollutants. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of a healthy diet
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 62
Participants
  baseline | 56
  post-study: number analyzed (Participants) | 56
  post-study | 48

18. Secondary Outcome: Knowledge of Which Foods Contain Phytonutrients
Description: Participants will be asked a question about which foods contain phytonutrients. Possible answers are meat, dairy, plant foods, all foods, or don't know. Data will be presented as the number of participants in each group that correctly identified plant foods.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 62
Participants
  baseline | 42
  post-study: number analyzed (Participants) | 56
  post-study | 37

19. Secondary Outcome: Knowledge of Environmental Pollutants
Description: Participants will be asked to identify environmental pollutants from a list. Possible answers are polychlorinated biphenyls (PCBs), mercury, nitrites, all of those, none of those, or don't know. Data will be presented as the number of participants in each group that correctly identified all of those.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group
Number analyzed (Participants) | 62
Participants
  baseline | 40
  post-study: number analyzed (Participants) | 56
  post-study | 36

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for this study.
Description: Adverse event data were not collected for this study.
Arm/Group | Walking Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT05002972/Prot_SAP_ICF_000.pdf